CLINICAL TRIAL: NCT03556241
Title: Perioperative Management of Patients With Pacemakers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: periop pacemaker
Record Dates: First submitted 2017-04-24; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Preoperative State; Presence of Pacemaker

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: No change group (Experimental): Case management consists keeping patient's current pacemaker mode during surgery
  Interventions: Device: Case management
- Control: Mode change group (No Intervention): Usual care consists changing pacemaker mode to VOO before surgery

INTERVENTIONS:
Device: Case management — Case management consists keeping patient's current pacemaker mode during surgery
  Arms: Intervention: No change group

SUMMARY:
Traditionally, when a patient who received permanent pacemaker undergoes surgery, physicians change pacemaker mode to DDD and recommend to use bipolar electrocautery to minimize electromagnetic interference. However, pacemaker function is improving and there's diverse suggestions for such situations. The investigators aimed to contemplate the necessity of perioperative pacemaker mode change. Patients with permanent pacemaker undergoing surgery are randomized into two groups by 1:1 ratio. No mode change is applied before surgery in case group and VOO is applied before surgery in control group. Perioperative adverse event would be compared in both groups.

DETAILED DESCRIPTION:
It has been more than 50 years after pacemaker device is developed. The subjects receiving permanent pacemaker has been increased and the number of patients with pacemaker undergoing surgery has been increased in company. However, in cases using electrocautery during surgery, there is possibility of malfunction of pacemaker due to electromagnetic interference. The factors associated with pacemaker malfunction during surgery have been reported; type of pacemaker, intrinsic heart rate, pacemaker dependency, type of electrocautery, position of generator, distance between generator/lead and electrocautery, duration and power of electrical energy. Conventionally, mode change to VOO before surgery and use of bipolar electrocautery are recommended before surgery but diverse suggestions regarding perioperative pacemaker mode change has been raised. The investigators aimed to contemplate the necessity of perioperative pacemaker mode change by prospective randomized trial. Patients with permanent pacemaker undergoing surgery are randomized into two groups by 1:1 ratio. No mode change is applied before surgery in the case group and VOO mode is applied before surgery in the control group. Exclusion criteria is thoracic surgery, 100% pacemaker dependency and unipolar pacing. The investigators will compare perioperative adverse events. The primary endpoint is asystole and the secondary endpoint is cardiac arrest, pacing inhibition, torsades de pointes and R on T.

ELIGIBILITY:
Inclusion Criteria:

* over 19 years old Patients undergoing surgery using electrocautery who received permanent pacemaker

Exclusion Criteria:

* Thoracic surgery (lung, esophagus, heart, breast) Totally pacemaker dependent patient. Unipolar pacing

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-02 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of asystole | Perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Seog Oh, MD,PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Seoul St Mary's Hospital, Seoul, Seo Ch-gu, South Korea